CLINICAL TRIAL: NCT04895358
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study of Pembrolizumab Plus Chemotherapy Versus Placebo Plus Chemotherapy for the Treatment of Chemotherapy-Candidate Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative (HR+/HER2-) Locally Recurrent Inoperable or Metastatic Breast Cancer (KEYNOTE-B49)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Chemotherapy Versus Placebo Plus Chemotherapy for HR+/HER2- Locally Recurrent Inoperable or Metastatic Breast Cancer (MK-3475-B49/KEYNOTE-B49)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-B49; MK-3475-B49 (Other: MSD); KEYNOTE-B49 (Other: MSD); 2023-506752-24 (Registry Identifier: EU CT); U1111-1294-3354 (Registry Identifier: UTN); jRCT2051210049 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); PHRR210721-003751 (Registry Identifier: Philippine Health Research Registry (PHRR)); 2020-005407-38 (EudraCT Number)
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms
Keywords: programmed cell death receptor 1 (PD-1, PD1); programmed cell death receptor ligand 1 (PD-L1, PDL1); programmed cell death receptor ligand 2 (PD-L2, PDL2); human epidermal growth factor 2 negative (HER2-); hormone receptor positive (HR+); estrogen receptor positive (ER+); progesterone receptor positive (PR+); metastatic; inoperable
MeSH Terms: conditions — Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body; Neoplasm Metastasis | interventions — pembrolizumab; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; liposomal doxorubicin; Capecitabine; Saline Solution; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Chemotherapy (Experimental): Participants receive pembrolizumab 200 mg administered by intravenous infusion (IV) on Day 1 of each 21-day cycle (Q3W) PLUS one of four chemotherapy regimens: 1) paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle (Q4W), 2) nab-paclitaxel 100 mg/m^2 IV on Days 1, 8, and 15 Q4W, 3) liposomal doxorubicin 50 mg/m^2 IV on Day 1 Q4W, OR 4) capecitabine 1000 mg/m^2 by oral administration (PO) twice a day (BID) on Days 1-14 Q3W for up to 35 administrations.
  Interventions: Biological: pembrolizumab; Drug: paclitaxel; Drug: nab-paclitaxel; Drug: liposomal doxorubicin; Drug: capecitabine
- Placebo + Chemotherapy (Active Comparator): Participants receive placebo (normal saline or dextrose) IV on Day 1 Q3W PLUS one of four chemotherapy regimens: 1) paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 Q4W, 2) nab-paclitaxel 100 mg/m^2 IV on Days 1, 8, and 15 Q4W, 3) liposomal doxorubicin 50 mg/m^2 IV on Day 1 Q4W, OR 4) capecitabine 1000 mg/m^2 PO BID on Days 1-14 Q3W for up to 35 administrations.
  Interventions: Drug: paclitaxel; Drug: nab-paclitaxel; Drug: liposomal doxorubicin; Drug: capecitabine; Drug: normal saline; Drug: dextrose

INTERVENTIONS:
Biological: pembrolizumab — Intravenous (IV) infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + Chemotherapy
Drug: paclitaxel — IV infusion
  Other Names: TAXOL®
Drug: nab-paclitaxel — IV infusion
  Other Names: ABRAXANE®
Drug: liposomal doxorubicin — IV infusion
  Other Names: DOXIL®
Drug: capecitabine — oral administration
  Other Names: XELODA®
Drug: normal saline — IV infusion
  Arms: Placebo + Chemotherapy
Drug: dextrose — IV infusion
  Arms: Placebo + Chemotherapy

SUMMARY:
The safety and efficacy of pembrolizumab plus the investigator's choice of chemotherapy will be assessed compared to placebo plus the investigator's choice of chemotherapy in the treatment of chemotherapy-candidate hormone receptor-positive, human epidermal growth factor receptor 2-negative (HR+/HER2-) locally recurrent inoperable or metastatic breast cancer.

The primary hypotheses are that the combination of pembrolizumab and chemotherapy is superior to placebo and chemotherapy in regards to Progression-Free Survival (PFS) in participants with programmed cell death-ligand 1 (PD-L1) combined positive score (CPS) ≥1.

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has locally recurrent inoperable or metastatic HR+/HER2- breast cancer, which has not been previously treated with cytotoxic chemotherapy in the noncurative setting
* Has progressed on prior endocrine therapy and is now a chemotherapy candidate, meeting the characteristics in regard to previous treatments of one of the following 4 groups:
* Group 1: Has progressed on 2 or more lines of endocrine therapy for advanced/metastatic HR+/HER2-disease, with at least given in combination with a Cyclin-dependent kinase 4/6 (CDK4/6) inhibitor. Prior treatment with mTOR and/or PI3-K inhibitors is allowed. OR
* GROUP 2a: Has progressed on 1 line of previous endocrine therapy for advanced/metastatic disease AND had a disease recurrence within 24 months of definitive surgery for the primary tumor and while on adjuvant endocrine therapy. Prior use of CDK4/6 inhibitors is required, either in the adjuvant and/or metastatic setting. Prior treatment with mTOR and/or PI3-K inhibitors is allowed. OR
* GROUP 2b: Has progressed within 12 months of starting 1 line of endocrine therapy with a CDK4/6 inhibitor for advanced/metastatic HR+/HER2- disease. OR
* GROUP 3: If no prior treatment with a CDK4/6 inhibitor, for advanced/metastatic disease and/or early stage disease (adjuvant), participants must have progressed within 6 months of starting 1 line of endocrine therapy with or without an mTOR or PI3-K inhibitor for metastatic disease AND had a relapse within 24 months of definitive surgery for primary tumor and while receiving adjuvant endocrine therapy.
* Has presented a documented radiographic disease progression (as assessed by the investigator and/or histology [biopsy or cytology] for participants presenting with new metastatic lesions) during or after the last administered endocrine therapy prior to entering the study.
* Is a chemotherapy candidate that meets the criteria specified in the protocol
* Provides a new or the last obtained core biopsy, preferably consisting of multiple cores, taken from a locally recurrent or a distant (metastatic) lesion not previously irradiated
* Has centrally confirmed PD-L1 CPS ≥1 and HR+ (estrogen receptor [ER] and/or progesterone receptor [PgR]) /HER2- breast cancer as defined by the most recent American Society of Clinical Oncology (ASCO)/(College of American Pathologists) CAP guidelines on most recent tumor biopsy
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 7 days prior to the first dose of study treatment
* Has adequate organ function within 10 days prior to the start of study
* Male participants must agree to the following during the treatment period and for at least 6 months after the last dose of chemotherapy: refrain from donating sperm PLUS either be abstinent from heterosexual intercourse as their preferred and usual lifestyle or use contraception and agree to use a male condom plus partner use of an additional contraceptive
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using a highly-effective contraceptive method during the treatment period and for at least 120 days after the last dose of pembrolizumab and 180 days after the last dose of chemotherapy (whichever occurs last), AND agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum) within 24 hours for urine or within 72 hours for serum before the first dose of study intervention
* Has measurable disease per RECIST 1.1 as assessed by the local site investigator/radiologist
* If receiving bisphosphonates or RANK ligand inhibitors, with stable doses for ≥4 weeks prior to the date of randomization, the participant may continue receiving this therapy during the study treatment. If participant needs to initiate these agents during the screening period, a bone scan to evaluate bone disease should be performed prior to randomization.
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks prior to the first dose of study intervention and have undetectable HBV viral load prior to randomization
* Participants with history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening

Exclusion Criteria:

* Has breast cancer amenable to treatment with curative intent
* Has a history or current evidence of any condition (e.g., transfusion-dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that is specifically contraindicated per the current locally-approved labeling, that might confound the results of the study, interfere with the participant's involvement for the full duration of the study, or is not in the best interest of the participant to be involved, in the opinion of the treating investigator
* Has significant cardiac disease, such as: history of myocardial infarction, acute coronary syndrome, coronary angioplasty/stenting/bypass within the last 6 months, congestive heart failure (CHF) New York Heart association (NYHA) Class II-IV, or history of CHF NYHA Class III or IV
* Has advanced/metastatic, symptomatic visceral spread at risk of rapidly evolving into life-threatening complications, such as lymphangitic lung metastases, bone marrow replacement, carcinomatous meningitis, significant symptomatic liver metastases, shortness of breath requiring supplemental oxygen, symptomatic pleural effusion requiring supplemental oxygen, symptomatic pericardial effusion, symptomatic peritoneal carcinomatosis, or the need to achieve rapid symptom control
* Has skin only disease
* Has a known germline BRCA mutation (deleterious or suspected deleterious) and has not received previous treatment with PARP inhibition. either in the adjuvant or metastatic setting (where available and not medically contraindicated). Single-agent PARP inhibitor therapy does not count as a line of endocrine therapy.
* Has received prior chemotherapy for locally recurrent inoperable or metastatic breast cancer
* Has received prior therapy with an anti- programmed cell death 1 (PD-1), anti- programmed cell death ligand 1 (PD-L1), or anti- programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137)
* Has received prior systemic anticancer therapy with other investigational agents within 4 weeks prior to randomization
* Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids.
* Has received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ excluding cancer in situ of bladder that have undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases
* Has diagnosed carcinomatous meningitis
* Has severe hypersensitivity to pembrolizumab and/or any of its excipients or has any hypersensitivity to the planned chemotherapy agent (paclitaxel, nab-paclitaxel, liposomal doxorubicin, or capecitabine) and/or any of their excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Has a known COVID-19 infection (symptomatic or asymptomatic)
* Has a known history of active tuberculosis (TB)
* Has a known psychiatric or substance abuse disorder including alcohol or drug dependency that would interfere with the participant's ability to cooperate with the requirements of the study
* Is breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days (or longer as specified by local institutional guidelines) after the last dose of study treatment
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2027-12-18 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With Combined Positive Score (CPS) ≥1 | Up to approximately 50 months
  PFS is defined as the time from randomization to the first documented disease progression (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The PFS in participants with a CPS of ≥1, as assessed by BICR, will be presented.

SECONDARY OUTCOMES:
Overall Survival (OS) in Participants With Combined Positive Score (CPS) ≥1 | Up to approximately 76 months
  OS is defined as the time from randomization to death due to any cause. OS for participants with a CPS of ≥1 will be presented.
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With Combined Positive Score (CPS) ≥10 | Up to approximately 76 months
  PFS is defined as the time from randomization to the first documented disease progression (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The PFS in participants with a CPS of ≥10, as assessed by BICR, will be presented.
OS in Participants With CPS ≥10 | Up to approximately 76 months
  OS is defined as the time from randomization to death due to any cause. OS for participants with a CPS of ≥10 will be presented.
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Investigator in Participants With Combined Positive Score (CPS) ≥10 | Up to approximately 76 months
  PFS is defined as the time from randomization to the first documented disease progression (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The PFS in participants with a CPS of ≥10, as assessed by investigator, will be presented.
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Investigator in Participants With Combined Positive Score (CPS) ≥1 | Up to approximately 76 months
  PFS is defined as the time from randomization to the first documented disease progression (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The PFS in participants with a CPS of ≥1, as assessed by investigator, will be presented.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With Combined Positive Score (CPS) ≥10 | Up to approximately 76 months
  ORR is defined as the percentage of participants in the analysis population who achieve confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. ORR for participants with a CPS of ≥10 will be presented.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With Combined Positive Score (CPS) ≥1 | Up to approximately 76 months
  ORR is defined as the percentage of participants in the analysis population who achieve confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. ORR for participants with a CPS of ≥1 will be presented.
Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With Combined Positive Score (CPS) ≥10 | Up to approximately 76 months
  DCR is defined as the percentage of participants who achieve Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions), or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD]) for at least 24 weeks. The percentage of participants who experience a confirmed CR, PR, or SD with a CPS of ≥10 will be presented.
Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With Combined Positive Score (CPS) ≥1 | Up to approximately 76 months
  DCR is defined as the percentage of participants who achieve Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions), or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD]) for at least 24 weeks. The percentage of participants who experience a confirmed CR, PR, or SD with a CPS of ≥1 will be presented.
Duration of Response (DOR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With Combined Positive Score (CPS) ≥10 | Up to approximately 76 months
  For participants who demonstrate CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the time from the first documented evidence of CR or PR until disease progression (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, or death from any cause, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. DOR for participants with a CPS of ≥10 will be presented.
Duration of Response (DOR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With Combined Positive Score (CPS) ≥1 | Up to approximately 76 months
  For participants who demonstrate CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the time from the first documented evidence of CR or PR until disease progression (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, or death from any cause, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. DOR for participants with a CPS of ≥1 will be presented.
Change From Baseline in Global Health Status/Quality of Life Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score will be presented in participants with a CPS of ≥10. A higher score indicates a better outcome.
Change From Baseline in Global Health Status/Quality of Life Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score will be presented in participants with a CPS of ≥1. A higher score indicates a better outcome.
Change From Baseline in Physical Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the physical functioning score will be presented in participants with a CPS of ≥10. A higher score indicates a better level of function.
Change From Baseline in Physical Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the physical functioning score will be presented in participants with a CPS of ≥1. A higher score indicates a better level of function.
Change From Baseline in Emotional Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 4 questions about their emotional functioning (Items 21-24) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the emotional functioning score will be presented in participants with a CPS of ≥10. A higher score indicates a better level of function.
Change From Baseline in Emotional Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 4 questions about their emotional functioning (Items 21-24) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the emotional functioning score will be presented in participants with a CPS of ≥1. A higher score indicates a better level of function.
Change From Baseline in Fatigue Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 3 questions about their fatigue (Items 10, 12, 18) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the fatigue score will be presented in participants with a CPS of ≥10. A lower score indicates a better outcome.
Change From Baseline in Fatigue Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 3 questions about their fatigue (Items 10, 12, 18) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the fatigue score will be presented in participants with a CPS of ≥1. A lower score indicates a better outcome.
Change From Baseline in Diarrhea Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire, including a single-item scale score for diarrhea (QLQ-C30 Item 17). For this item, individual responses to the question "Have you had diarrhea?" are given on a 4-point scale (1=Not at all; 4=Very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the diarrhea score will be presented in participants with a CPS of ≥10. A lower score indicates a better outcome.
Change From Baseline in Diarrhea Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Baseline and up to approximately 76 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire, including a single-item scale score for diarrhea (QLQ-C30 Item 17). For this item, individual responses to the question "Have you had diarrhea?" are given on a 4-point scale (1=Not at all; 4=Very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the diarrhea score will be presented in participants with a CPS of ≥1. A lower score indicates a better outcome.
Time to Deterioration (TTD) in Global Health Status/Quality of Life Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in Global Health Status (GHS; EORTC QLQ-C30 Item 29) & Quality of Life (QoL; EORTC QLQ-C30 Item 30) combined score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in GHS and QoL combined score, will be presented in participants with a CPS of ≥10. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Global Health Status/Quality of Life Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in Global Health Status (GHS; EORTC QLQ-C30 Item 29) & Quality of Life (QoL; EORTC QLQ-C30 Item 30) combined score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in GHS and QoL combined score, will be presented in participants with a CPS of ≥1. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Physical Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in physical functioning score (EORTC QLQ-C30 Items 1-5). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in physical functioning score, will be presented in participants with a CPS of ≥10. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Physical Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in physical functioning score (EORTC QLQ-C30 Items 1-5). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in physical functioning score, will be presented in participants with a CPS of ≥1. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Diarrhea Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in diarrhea score (EORTC QLQ-C30 Item 17). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in diarrhea score, will be presented in participants with a CPS of ≥10. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Emotional Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in emotional functioning score (EORTC QLQ-C30 Items 21-24). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in emotional functioning score, will be presented in participants with a CPS of ≥10. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Emotional Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in emotional functioning score (EORTC QLQ-C30 Items 21-24). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in emotional functioning score, will be presented in participants with a CPS of ≥1. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Fatigue Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥10 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in fatigue score (EORTC QLQ-C30 Items 10, 12, 18). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in fatigue score, will be presented in participants with a CPS of ≥10. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Fatigue Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in fatigue score (EORTC QLQ-C30 Items 10, 12, 18). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in fatigue score, will be presented in participants with a CPS of ≥1. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in Diarrhea Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in Participants with CPS ≥1 | Up to approximately 76 months
  TTD is defined as the time to the first onset of a ≥10-point deterioration (decrease) from baseline in diarrhea score (EORTC QLQ-C30 Item 17). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point deterioration (decrease) from baseline in diarrhea score, will be presented in participants with a CPS of ≥1. A longer TTD indicates a better outcome.
Percentage of Participants who Experience an Adverse Event (AE) | Up to approximately 76 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experience one or more adverse events will be presented.
Percentage of Participants who Discontinue Study Drug due to an AE | Up to approximately 76 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinue study treatment due to an adverse event will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (256):
- United States (41):
  - University of Alabama at Birmingham-Medicine ( Site 0065), Birmingham, Alabama
  - Arizona Oncology Associates-Arizona Oncology ( Site 0049), Tucson, Arizona
  - Pacific Cancer Care ( Site 0023), Monterey, California
  - UCSF Medical Center at Mission Bay ( Site 0043), San Francisco, California
  - Georgetown University Medical Center-Department of Medicine and Oncology ( Site 0026), Washington D.C., District of Columbia
  - MedStar Washington Hospital Center ( Site 0063), Washington D.C., District of Columbia
  - Baptist MD Anderson Cancer Center ( Site 0013), Jacksonville, Florida
  - Miami Cancer Institute at Baptist Health, Inc. ( Site 0070), Miami, Florida
  - Miami Cancer Institute - Plantation ( Site 0076), Plantation, Florida
  - University Cancer & Blood Center, LLC ( Site 0032), Athens, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 0028), Marietta, Georgia
  - University of Illinois at Chicago ( Site 0061), Chicago, Illinois
  - Edward-Elmhurst Healthcare, Elmhurst Hospital-Nancy W. Knowles Cancer Center ( Site 0067), Elmhurst, Illinois
  - Edward-Elmhurst Healthcare, Edward Hospital-Edward Cancer Center ( Site 0066), Naperville, Illinois
  - Edward-Elmhurst Healthcare, Edward Hospital - Plainfield-Edward Cancer Center - Plainfield ( Site 00, Plainfield, Illinois
  - Orchard Healthcare Research Inc. ( Site 0037), Skokie, Illinois
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0071), Fort Wayne, Indiana
  - McFarland Clinic, PC ( Site 0041), Ames, Iowa
  - Louisiana State University Health Sciences Shreveport ( Site 0072), Shreveport, Louisiana
  - CHRISTUS Highland-Oncology Research ( Site 0073), Shreveport, Louisiana
  - New England Cancer Specialists ( Site 0007), Scarborough, Maine
  - Greater Baltimore Medical Center-Medical Oncology/Hematology ( Site 0062), Baltimore, Maryland
  - MFSMC-HJWCI ( Site 0064), Baltimore, Maryland
  - MedStar Good Samaritan Hospital-Oncology Research ( Site 0069), Baltimore, Maryland
  - University of Massachusetts Medical School-Division of Hematology/Oncology ( Site 0052), Worcester, Massachusetts
  - Henry Ford Hospital ( Site 0003), Detroit, Michigan
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0009), Omaha, Nebraska
  - Broome Oncology ( Site 0018), Johnson City, New York
  - Hematology Oncology Associates of Rockland ( Site 0044), Nyack, New York
  - Waverly Hematology Oncology ( Site 0015), Cary, North Carolina
  - Sanford Fargo Medical Center ( Site 0040), Fargo, North Dakota
  - Providence Portland Medical Center ( Site 0038), Portland, Oregon
  - Oregon Health and Science University ( Site 0031), Portland, Oregon
  - St Francis Cancer Center ( Site 0058), Greenville, South Carolina
  - Sanford Cancer Center ( Site 0021), Sioux Falls, South Dakota
  - University of Tennessee Medical Center ( Site 0039), Knoxville, Tennessee
  - Bon Secours St. Francis Medical Center-Oncology Research ( Site 0020), Midlothian, Virginia
  - Kadlec Clinic Hematology and Oncology ( Site 0055), Kennewick, Washington
  - Medical Oncology Associates, PS ( Site 0010), Spokane, Washington
  - Northwest Medical Specialties, PLLC ( Site 0008), Tacoma, Washington
  - North Star Lodge ( Site 0035), Yakima, Washington
- Argentina (11):
  - Centro de Oncología e Investigación de Buenos Aires ( Site 0400), Berazategui, Buenos Aires
  - Hospital Británico de Buenos Aires-Oncology ( Site 0404), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0412), Mar del Plata, Buenos Aires
  - Hospital Aleman-Oncology ( Site 0402), Buenos Aires, Buenos Aires F.D.
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC) ( Site 0403), Buenos Aires, Buenos Aires F.D.
  - Sanatorio de La Mujer ( Site 0405), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 0407), Rosario, Santa Fe Province
  - Instituto de Oncología de Rosario ( Site 0401), Rosario, Santa Fe Province
  - Hospital Italiano de Córdoba ( Site 0409), Córdoba
  - Fundación CEMAIC ( Site 0410), Córdoba
  - Instituto San Marcos ( Site 0408), San Juan
- Australia (4):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 2102), Macquarie Park, New South Wales
  - Westmead Hospital-Department of Medical Oncology ( Site 2101), Westmead, New South Wales
  - Frankston Hospital-Oncology and Haematology ( Site 2103), Frankston, Victoria
  - Breast Cancer Research Centre-WA ( Site 2104), Nedlands, Western Australia
- Austria (5):
  - Landesklinikum Wiener Neustadt-Innere Medizin, Hämatologie und internistische Onkologie ( Site 1604), Wiener Neustadt, Lower Austria
  - Medizinische Universität Graz-Innere Medizin Klin. Abt. Onkologie ( Site 1609), Graz, Styria
  - Medizinische Universitaet Innsbruck ( Site 1602), Innsbruck, Tyrol
  - Medizinische Universität Wien ( Site 1601), Vienna, Vienna
  - Uniklinikum Salzburg-Universitätsklinik für Innere Medizin III der PMU mit Hämatologie, internistis, Salzburg
- Brazil (6):
  - Hospital de Câncer de Recife ( Site 0211), Recife, Pernambuco
  - Instituto de Oncologia Saint Gallen ( Site 0206), Santa Cruz do Sul, Rio Grande do Sul
  - Clínica de Oncologia Reichow ( Site 0210), Blumenau, Santa Catarina
  - YNOVA Pesquisa Clínica ( Site 0203), Florianópolis, Santa Catarina
  - Instituto Nacional de Câncer - INCA-Pesquisa Clinica HC3 ( Site 0208), Rio de Janeiro
  - Instituto de Educação, Pesquisa e Gestão em Saúde ( Site 0202), Rio de Janeiro
- Canada (7):
  - Tom Baker Cancer Center ( Site 0107), Calgary, Alberta
  - North York General Hospital ( Site 0108), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0101), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal ( Site 0105), Montreal, Quebec
  - Jewish General Hospital ( Site 0110), Montreal, Quebec
  - Hopital Du Saint-Sacrement ( Site 0109), Québec, Quebec
  - Centre integre universitaire de sante et de services sociaux de la Mauricie-et-du-centre-du-quebec (, Trois-Rivières, Quebec
- Chile (6):
  - FALP ( Site 0501), Santiago, Region M. de Santiago
  - Oncovida ( Site 0514), Santiago, Region M. de Santiago
  - Clínica RedSalud Vitacura ( Site 0515), Santiago, Region M. de Santiago
  - Instituto Nacional del Cancer-CR Investigación ( Site 0511), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0500), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0513), Temuco, Región de la Araucanía
- China (27):
  - Anhui Cancer Hospital-medical oncology ( Site 2632), Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science ( Site 2635), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Department of Breast Cancer ( Site 2605), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-Medical Oncology ( Site 2610), Beijing, Beijing Municipality
  - The First Affiliated hospital of Xiamen University-Breast Surgery ( Site 2613), Xiamen, Fujian
  - The First People's Hospital of Foshan-Oncology Department of Breast Cancer ( Site 2620), Foshan, Guangdong
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE-oncology breast ( Site 2616), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University-Breast Oncology Center ( Site 2641), Guangzhou, Guangdong
  - Peking University Shenzhen Hospital-Oncology Department ( Site 2601), Shenzhen, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital-Oncology Dept. of Breast and Bone Soft Tissue (, Nanning, Guangxi
  - Henan Cancer Hospital-Galactophore Department ( Site 2615), Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center-Cancer Center ( Site 2629), Wuhan, Hubei
  - Xiangya Hospital Central South University-Breast department ( Site 2621), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 2608), Changsha, Hunan
  - Jiangsu provincial people's hospital-Oncology Department ( Site 2607), Nanjing, Jiangsu
  - The Third Hospital of Nanchang-Oncology Dept ( Site 2628), Nanchang, Jiangxi
  - Jilin Cancer Hospital-oncology department ( Site 2619), Changchun, Jilin
  - The First Affiliated Hospital of Xian Jiaotong University wa-Oncology ( Site 2604), Xi'an, Shaanxi
  - Shandong Cancer Hospital-Breast surgery ( Site 2623), Jinan, Shandong
  - Fudan University Shanghai Cancer Center-Oncology ( Site 2600), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiao Tong University School of Medicine-Breast surgery ( Site 2626), Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University-Head and Neck Oncology ( Site 2630), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital-Department of Breast Cancer ( Site 2612), Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi-galactophore department ( Site 2624), Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital-Breast Oncology ( Site 2622), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 2636), Linhai, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Thyroid and breast surgery ( Site 2625), Wenzhou, Zhejiang
- Colombia (6):
  - Fundación Colombiana de Cancerología Clínica Vida ( Site 0605), Medellín, Antioquia
  - Instituto de Cancerología-Oncology ( Site 0606), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 0601), Barranquilla, Atlántico
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 0607), Bogotá, Bogota D.C.
  - Sociedad De Oncologia Y Hematologia Del Cesar-Oncology ( Site 0603), Valledupar, Cesar Department
  - Oncomedica S.A.-Oncomedica S.A ( Site 0604), Montería, Departamento de Córdoba
- France (14):
  - CENTRE LEON BERARD ( Site 0919), Lyon, Auvergne-Rhône-Alpes
  - Institut Paoli-Calmettes ( Site 0913), Marseille, Bouches-du-Rhone
  - Centre François Baclesse ( Site 0920), Caen, Calvados
  - CHU Besançon ( Site 0918), Besançon, Franche-Comte
  - Institut Claudius Regaud ( Site 0902), Toulouse, Haute-Garonne
  - Centre de Cancérologie du Grand Montpellier ( Site 0912), Montpellier, Languedoc-Roussillon
  - Institut de Cancérologie de l'Ouest ( Site 0907), Saint-Herblain, Loire-Atlantique
  - Institut de Cancérologie de l'Ouest ( Site 0915), Angers, Maine-et-Loire
  - Centre Oscar Lambret ( Site 0921), Lille, Nord
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne ( Site 0901), Clermont-Ferrand, Puy-de-Dome
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen ( Site 0904), Rouen, Seine-Maritime
  - Centre Hospitalier Universitaire de Poitiers-Pôle régional de cancérologie ( Site 0922), Poitiers, Vienne
  - Institut Curie ( Site 0900), Paris
  - Gustave Roussy ( Site 0914), Villejuif, Île-de-France Region
- Germany (6):
  - Universitaetsklinikum Erlangen-Klinik für Gynäkologie und Geburtshilfe ( Site 1202), Erlangen, Bavaria
  - Gynaekologisches Zentrum Bonn ( Site 1201), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf-Klinik für Frauenheilkunde & Geburtshilfe ( Site 1204), Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung-Klinike für Senologie/ Brustzentrum ( Site 1200, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Frauenheilkunde und Gebur, Dresden, Saxony
  - Vivantes Klinikum Am Urban-Haematologie und Onkologie ( Site 1203), Berlin
- Greece (5):
  - General Hospital of Athens Laiko-First Department of Internal Medicine ( Site 0305), Athens, Attica
  - Alexandra Hospital-ONCOLGOY DEPT. ( Site 0302), Athens, Attica
  - Hygeia Hospital-3rd Oncology Department ( Site 0304), Marousi, Attica
  - University General Hospital of Heraklion-Internal Medicine-Oncology ( Site 0303), Heraklion, Irakleio
  - Euromedica General Clinic Thessaloniki-Oncology Unit ( Site 0301), Thessaloniki
- Guatemala (4):
  - CELAN,S.A ( Site 0151), Guatemala City
  - Gastrosoluciones ( Site 0156), Guatemala City
  - INTEGRA Cancer Institute ( Site 0155), Guatemala City
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 0154), Quetzaltenango
- Hungary (3):
  - Pécsi Tudományegyetem Klinikai Központ-Onkoterápiás Intézet ( Site 2807), Pécs, Baranya
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 2804), Kecskemét, Bács-Kiskun county
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Onkoterapias Klinika ( Site 2805), Szeged, Csongrád megye
- Ireland (2):
  - St. James's Hospital ( Site 1530), Dublin
  - St. Vincent's University Hospital-Medical Oncology Research Department ( Site 1531), Dublin
- Israel (5):
  - Assuta Ashdod Medical Center ( Site 1703), Ashdod
  - Soroka Medical Center-Oncology ( Site 1702), Beersheba
  - Bnai Zion Medical Center-Oncology ( Site 1704), Haifa
  - Sheba Medical Center-ONCOLOGY ( Site 1700), Ramat Gan
  - Sourasky Medical Center-Oncology ( Site 1701), Tel Aviv
- Italy (9):
  - Fondazione Policlinico Universitario Agostino Gemelli-Medical Oncology ( Site 1113), Rome, Lazio
  - Ospedale San Raffaele-Oncologia Medica ( Site 1110), Milan, Lombardy
  - Ospedale San Gerardo-ASST Monza-Research Unit Phase 1 ( Site 1115), Monza, Lombardy
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1114), Rozzano, Milano
  - Instituto Tumori Giovanni Paolo II-ONCOLOGIA MEDICA ( Site 1112), Bari
  - Ospedale Cannizzaro ( Site 1118), Catania
  - Istituto Europeo di Oncologia IRCCS-Divisione di Senologia Medica ( Site 1111), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1116), Napoli
  - Istituto Oncologico Veneto IRCCS ( Site 1117), Padua
- Japan (12):
  - Hyogo Medical University Hospital ( Site 2201), Nishinomiya, Hyōgo
  - St. Marianna University School of Medicine Hospital ( Site 2205), Kawasaki, Kanagawa
  - Kitasato University Hospital ( Site 2204), Sagamihara, Kanagawa
  - Osaka University Hospital ( Site 2211), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 2208), Hidaka, Saitama
  - Tokyo Medical University Hospital ( Site 2206), Shinjuku-ku, Tokyo
  - Chiba University Hospital ( Site 2212), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 2209), Fukuoka
  - Fukushima Medical University ( Site 2200), Fukushima
  - Kumamoto University ( Site 2203), Kumamoto
  - St. Luke's International Hospital ( Site 2207), Tokyo
  - Juntendo University Hospital ( Site 2210), Tokyo
- Malaysia (5):
  - University Malaya Medical Centre ( Site 2505), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 2504), George Town, Pulau Pinang
  - Sarawak General Hospital-Radiotherapy Unit ( Site 2501), Kuching, Sarawak
  - Hospital Kuala Lumpur-Radiotherapy and Oncology ( Site 2506), Kuala Lumpur
  - Pantai Hospital Kuala Lumpur-Cancer Centre ( Site 2503), Kuala Lumpur
- Mexico (5):
  - Hospital Civil Fray Antonio Alcalde-Oncology ( Site 0262), Guadalajara, Jalisco
  - Samadhi Centro Oncológico ( Site 0258), Mexico City, Mexico City
  - Filios Alta Medicina ( Site 0253), Monterrey, Nuevo León
  - Centro Estatal de Cancerologia-Investigación ( Site 0256), Chihuahua City
  - Centro de Investigacion Clinica de Oaxaca ( Site 0252), Oaxaca City
- Netherlands (9):
  - Radboudumc-Medical Oncology ( Site 1360), Nijmegen, Gelderland
  - Maastricht UMC+-Medical Oncology ( Site 1353), Maastricht, Limburg
  - Jeroen Bosch Hospital ( Site 1359), 's-Hertogenbosch, North Brabant
  - Elisabeth-TweeSteden Ziekenhuis-Internal Medicine ( Site 1357), Tilburg, North Brabant
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL) ( Site 1351), Amsterdam, North Holland
  - Leids Universitair Medisch Centrum-Medical Oncology ( Site 1356), Leiden, South Holland
  - Haaglanden MC - locatie Antoniushove-Medical oncology ( Site 1355), Leidschendam, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Vlietland ( Site 1354), Schiedam, South Holland
  - Meander Medisch Centrum ( Site 1358), Amersfoort, Utrecht
- Philippines (2):
  - East Avenue Medical Center ( Site 0802), Quezon City, National Capital Region
  - CARDINAL SANTOS MEDICAL CENTER-Research Room ( Site 0800), San Juan City, National Capital Region
- Poland (12):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1813), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow ( Site 1809), Krakow, Lesser Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 1818), Siedlce, Masovian Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 1820), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Piersi i Chirurgii (, Warsaw, Masovian Voivodeship
  - Lux med onkologia sp. z o.o. ( Site 1808), Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny-Klinika Onkologii ( Site 1803), Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Onkologiczny-BREAST CANCER ( Site 1821), Wieliszew, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1819), Przemyśl, Podkarpackie Voivodeship
  - Bialostockie Centrum Onkologii-Oddzial Onkologii Klinicznej ( Site 1812), Bialystok, Podlaskie Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach-Breast Unit ( Site 1811), Gliwice, Silesian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 1815), Koszalin, West Pomeranian Voivodeship
- Portugal (5):
  - Champalimaud Foundation ( Site 1006), Lisbon, Lisbon District
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E. - Hospital de Santa Maria ( Site 1004), Lisbon, Lisbon District
  - UNIDADE LOCAL DE SAUDE DE MATOSINHOS ( Site 1007), Matosinhos Municipality, Porto District
  - Centro Hospitalar do Porto - Hospital de Santo António-Oncology Service ( Site 1003), Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 1005), Porto
- Romania (5):
  - Cardiomed SRL Cluj-Napoca ( Site 2902), Cluj-Napoca, Cluj
  - Institutul Oncologic-Day Hospital Unit ( Site 2905), Cluj-Napoca, Cluj
  - Centrul de Oncologie "Sfântul Nectarie"-Medical Oncology ( Site 2901), Craiova, Dolj
  - Oncopremium Team-Oncology ( Site 2903), Baia Mare, Maramureş
  - Sigmedical Services SRL ( Site 2904), Suceava
- Russia (9):
  - Arkhangelsk Clinical Oncological Dispensary-Chemotherapy department ( Site 1902), Arkhangelsk, Arkhangelskaya oblast
  - Moscow Clinical Research Center-Chemotherapy department ( Site 1903), Moscow, Moscow
  - Fed State Budgetary Inst N.N. Blokhin Med Center of Oncology MHRF ( Site 1901), Moscow, Moscow
  - Central Clinical Hospital of the Presidential Administrative Department ( Site 1904), Moscow, Moscow
  - Podolsk Regional Clinical Hospital ( Site 1907), Podolsk, Moscow Oblast
  - Nizhegorodsky Regional Oncology Dispensary-chemotherapy ( Site 1912), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Ryazan Regional Clinical Oncology Center-Oncology #1 ( Site 1906), Ryazan, Ryazan Oblast
  - St. Petersburg Clinical Hospital of Russian Academy Of Sciences-Medical Oncology ( Site 1905), Saint Petersburg, Sankt-Peterburg
  - N.N.Petrov Research Institute of Oncology ( Site 1900), Saint Petersburg, Sankt-Peterburg
- South Korea (6):
  - National Cancer Center-Center for Breast Cancer ( Site 2404), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 2406), Seongnam, Kyonggi-do
  - Seoul National University Hospital-Internal Medicine ( Site 2403), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 2400), Seoul
  - Asan Medical Center ( Site 2402), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 2401), Seoul
- Spain (5):
  - Hospital Quiron Barcelona ( Site 1326), Barcelona, Catalonia
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 1323), Pozuelo de Alarcón, Madrid
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON ( Site 1333), Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 1320), Madrid, Madrid, Comunidad de
  - Fundación Instituto Valenciano de Oncología-Oncologico ( Site 1332), Valencia, Valenciana, Comunitat
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna-Tema Cancer - ME Bröst- endokrina tumörer och sarkom ( Site 1, Stockholm, Stockholm County
  - Södra Älvsborg Sjukhus ( Site 1406), Borås, Västra Götaland County
- Turkey (Türkiye) (11):
  - Ege University Medicine of Faculty ( Site 2004), Bornova, İzmir
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 2016), Izmir, Karsiyaka, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center ( Site 2013), Adana
  - Hacettepe Universitesi-oncology hospital ( Site 2000), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 2002), Ankara
  - Gazi Universitesi-Oncology ( Site 2010), Ankara
  - ANKARA ŞEHİR HASTANESİ-Medical Oncology ( Site 2014), Ankara
  - Akdeniz Universitesi Hastanesi-Medical Oncology ( Site 2009), Antalya
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 2012), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2005), Istanbul
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi Eğitim ve Araştırma Hastanesi-Medical Oncology Department, Malatya
- United Kingdom (7):
  - The Royal Cornwall Hospital ( Site 1507), Truro, Cornwall
  - Leicester Royal Infirmary-HOPE Clinical Trials Unit ( Site 1502), Leicester, England
  - St Bartholomew's Hospital ( Site 1508), London, England
  - The Christie ( Site 1510), Manchester, England
  - Blackpool Victoria Hospital ( Site 1503), Blackpool, Lancashire
  - Guy's & St Thomas' NHS Foundation Trust ( Site 1501), London, London, City of
  - North West Cancer Centre ( Site 1511), Londonderry, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26157&tenant=MT_MSD_9011